CLINICAL TRIAL: NCT06798805
Title: Unraveling the Role of Extracellular Vesicles-driven Senescence in Myeloproliferative Neoplasms
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: EVs-Sene; FIN-RER_BU_2020_29 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2024-12-30; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-12

CONDITIONS: Essential Thrombocythemia (ET); Myelofibrosis (MF); Polycythemia Vera (PV)
MeSH Terms: conditions — Thrombocythemia, Essential; Primary Myelofibrosis; Polycythemia Vera

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and mononuclear cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In this study the aim is to investigate the pathogenetic role of extracellular vesicles and senescence in Myeloproliferative Neoplasms. In particular, the goal of this project is to identify possible EV-based biomarkers of senescence according to gender, which are disease-specific, biology-related, and predictive of short-term outcome in terms of Event-Free Survival and to define personalized targets for new therapeutic approaches.

DETAILED DESCRIPTION:
This is a 3-year multi-centre prospective in vitro study. 120 patients with MPN (ET (n=45), PV (n=45), and MF (n=30)) will be enrolled for a period of 22 months. Follow-up: 12 months. Patients (ET=Group A; PV=Group B; MF=Group C) will be enrolled at the Complex Operative Unit of Haematology-IRCCS Azienda Ospedaliero-Universitaria di Bologna and at the Haematology Centres of Reggio Emilia, Brescia, Meldola, and Ravenna. Peripheral blood samples from patients with ET, PV, and MF (Group A-C; 40 ml) and/or bone marrow samples from patients with ET and PV (Group A, B; 5 ml) will be collected at diagnosis as part of normal clinical practice. The samples will be analysed at the Complex Operative Unit of Haematology-IRCCS Azienda Ospedaliero-Universitaria di Bologna in collaboration with the Istituto Romagnolo per lo Studio dei Tumori 'Dino Amadori' - IRST IRCCS (analysis of EV size and concentration) and with the University of Perugia (analysis of EV lipid cargo). The data analysis will be carried out in collaboration with the Department of Physics and Astronomy of the University of Bologna.

ELIGIBILITY:
Inclusion criteria for patients:

* age ≥ 18 years.
* patients with WHO2017-defined diagnosis of Myeloproliferative Neoplasms.
* patients at first diagnosis.
* Informed consent signed.

Exclusion criteria for patients:

- patients with concomitant second neoplasia

Inclusion criteria for Healthy Donors:

* age ≥ 18 years.
* Informed consent signed.

Exclusion criteria for Healthy Donors:

- Healthy Donors with neoplasia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Myeloproliferative Neoplasms (Essential Thrombocythemia, Polycythemia Vera, Myelofibrosis) will be enrolled over a 28 months period. Follow-up 1 year.
  As a control, sex/age matched Healthy Donors will be enrolled among volunteers of a no profit organization called AIL Bologna.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Plasma extracellular vesicle characterization | 2 years
  Comparison of concentration (particles/mL), phenotype, and cargo between extracellular vesicles from patients and healthy donors.
Validation of extracellular vesicles as biomarker | 2 years
  Correlation of extracellular vesicles' characterization data with markers of disease aggressiveness.

SECONDARY OUTCOMES:
Cell culture-derived extracellular vesicle characterization | 2 years
  Comparison of the phenotype of extracellular vesicles derived from the supernatant of selected immune cells cultured in the presence or absence of inflammatory factors.
Extracellular vesicle-mediated senescence | 1 years
  Comparison of senescence biomarkers (such as p16 and p21) in selected immune cells from healthy donors in the presence or absence of extracellular vesicles from patients or healthy donors.

OTHER OUTCOMES:
Validation of extracellular vesicles as biomarker | 1 years
  Development of an integrated analysis of clinical data and extracellular vesicle-based scenescence biomarkers to allow the identification of a short-term prognostic index in Myeloproliferative Neoplasm patients.

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Catani, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (5):
- Italy (5):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna
  - ASST Spedali Civili di Brescia, Brescia, BS
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori- IRST, Meldola, FC
  - Ospedale S.Maria delle Croci, Ravenna, RA
  - Arcispedale S. Maria Nuova - IRCCS, Reggio Emilia, RE